CLINICAL TRIAL: NCT04835441
Title: A Randomized, Double-blind, Placebo-controlled Study of ALPN-101 in Systemic Lupus Erythematosus
Brief Title: ALPN-101 (Acazicolcept) in Systemic Lupus Erythematosus
Acronym: Synergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alpine Immune Sciences Inc, A Subsidiary of Vertex (Industry)
Responsible Party: Sponsor
Organization: Alpine Immune Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIS-A03
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CD28; ICOS; Autoimmune disease; Immune system disease; Immunosuppressive agent
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Immune System Diseases | interventions — ALPN-101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALPN-101 (Acazicolcept) (Experimental): Participants received a weight-based dose of 3 milligrams/kilogram (mg/kg) ALPN-101 once every 2 weeks (Q2W) up to 24 weeks.
  Interventions: Drug: ALPN-101
- Placebo (Placebo Comparator): Participants received placebo matched to ALPN-101 up to 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALPN-101 — Intravenous infusion via an infusion pump.
  Other Names: Acazicolcept
  Arms: ALPN-101 (Acazicolcept)
Drug: Placebo — Intravenous infusion via an infusion pump.
  Arms: Placebo

SUMMARY:
This is Phase 2, multinational, randomized, blinded study to evaluate the safety, tolerability, efficacy, immunogenicity, pharmacokinetics and pharmacodynamics of ALPN-101 (acazicolcept) in adults with moderate to severe active systemic lupus erythematosus (SLE)

ELIGIBILITY:
Key Inclusion Criteria Summary

* SLE onset ≥ 6 months prior to Screening
* Positive ANA and/or elevated anti-dsDNA and/or elevated anti-Smith antibody test
* Active lupus at Screening and Baseline, as defined per-protocol and confirmed by the study's medical monitor, including a SLEDAI score at Screening of ≥ 6 and a clinical score at Baseline of ≥ 4
* Standard lupus medications must be stable prior to Screening

Key Exclusion Criteria Summary:

* Life-threatening or organ system-threatening lupus activity that is anticipated to require increased treatment during the study
* Proteinuria consistent with nephrotic syndrome
* Active lupus-related neuropsychiatric disease
* Drug-induced lupus
* Recent or serious ongoing infection; risk or history of serious infection
* Receipt of live vaccination within 8 weeks of Day 1, or expected to require live vaccination during the study
* Prior diagnosis of, or fulfills diagnostic criteria for, another rheumatic disease that overlaps with lupus or another autoimmune or inflammatory disease that may confound clinical assessments or increase subject risk in the study
* Diagnosis of, or fulfills diagnostic criteria for fibromyalgia
* Functional class IV
* Serious lupus disease activity, which warrants immediate immunosuppressive therapy not appropriate for the study or which makes the possibility of receiving placebo or investigational agent an inappropriate risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (29):
  - Investigational Site (107), Anniston, Alabama
  - Investigational Site (189), Phoenix, Arizona
  - Investigational Site (155), Los Angeles, California
  - Investigational Site (109), San Diego, California
  - Investigational Site (169), Santa Barbara, California
  - Investigational Site (106), DeBary, Florida
  - Investigational Site (120), Hialeah, Florida
  - Investigational Sites (134), Miami, Florida
  - Investigational Site (152), Ormond Beach, Florida
  - Investigational Site (133), Plantation, Florida
  - Investigational Site (190), Tamarac, Florida
  - Investigational Site (163), Tampa, Florida
  - Investigational Site (173), Idaho Falls, Idaho
  - Investigational Site (156), Skokie, Illinois
  - Investigational Site (138), Grand Blanc, Michigan
  - Investigational Site (164), Las Vegas, Nevada
  - Investigational Site (175), Brooklyn, New York
  - Investigational Site (115), Manhasset, New York
  - Investigational Site (179), Charlotte, North Carolina
  - Investigational Site (112), Crossville, Tennessee
  - Investigational Site (186), Memphis, Tennessee
  - Investigational Site (171), Baytown, Texas
  - Investigational Site (143), Bellaire, Texas
  - Investigational Site (118), Colleyville, Texas
  - Investigational Site (166), Fort Worth, Texas
  - Investigational Site (121), Houston, Texas
  - Investigational Site (104), Mesquite, Texas
  - Investigational Site (162), San Antonio, Texas
  - Investigational Site (127), San Antonio, Texas
- France (3):
  - Investigational Site (149), Marseille
  - Investigational Site (128), Paris
  - Investigational Site (161), Paris
- Hungary (3):
  - Investigational Site (181), Budapest
  - Investigational Site (180), Gyula
  - Investigational Site (183), Székesfehérvár
- Poland (5):
  - Investigational Site (160), Elblag
  - Investigational Site (110), Krakow
  - Investigational Site (108), Poznan
  - Investigational Site (119), Poznan
  - Investigational Site (165), Wroclaw
- Puerto Rico (2):
  - Investigational Site (191), Caguas
  - Investigational Site (187), San Juan
- Spain (2):
  - Investigational Site (137), A Coruña
  - Investigational Site (139), Seville
- Taiwan (2):
  - Investigational Site (184), Taichung
  - Investigational Site (182), Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in participants with active systemic lupus erythematosus (SLE) aged 18 years and older.
Period: Overall Study
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Started | 38 | 38
Completed | 33 | 32
Not Completed | 5 | 6
Not completed — Physician Decision | 4 | 4
Not completed — Other | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- ALPN-101 (Acazicolcept): Participants received a weight-based dose of 3mg/kg ALPN-101 Q2W up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | ALPN-101 (Acazicolcept) | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (11.20) | 47.8 (11.08) | 48.3 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 23 | 47
  Black or African American | 12 | 11 | 23
  Other Asian | 1 | 2 | 3
  American Indian or Alaska Native | 0 | 1 | 1
  East Asian | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Safety follow-up (up to 28 weeks)
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 38 | 38
Participants
  Participants with TEAEs | 23 | 24
  Participants with SAEs | 2 | 2

2. Primary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus (SLE) Responder Index (SRI)-4
Description: The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLE Disease Activity Index 2000 (SLEDAI-2K), the British Isles Lupus Assessment Group (BILAG) 2004 Index, and the Physician's Global Assessment (PGA). Participants classified as responder if they met all of the following criteria: 1) ≥ 4-point reduction in the SLEDAI-2K total score; 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B) compared with baseline; and 3) No worsening from baseline in participants' lupus disease activity (i.e., increase of ≥0.3 0 on a 3-point scale) in PGA. The SLEDAI-2K total score falls between 0 and 105, with higher scores representing increased disease activity. SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). BILAG: assesses disease extent, severity (range: A[severe] to E[no disease]). PGA: assesses worsening in participant's general health.
Time Frame: At Day 169
Population: Modified intent-to-treat population (mITT), includes all randomized participants who received any amount of study drug and have completed at least one post-baseline disease assessment. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
percentage of participants | 27 | 46
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.107, Cochran-Mantel-Haenszel

3. Primary Outcome: Percentage of Participants Achieving a British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) Response
Description: The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and Physician's Global Assessment (PGA). BICLA response is defined as: 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [mild disease] scores falling to C [Stable and mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4) ≤ 10% deterioration in PGA score. The PGA is measured on a 0 to 100 mm scale with score 0 indicates No Disease Activity and score 100 indicates the most Severe Disease Activity.
Time Frame: At Day 169
Population: mITT includes all randomized participants who received any amount of study drug and have completed at least one post-baseline disease assessment. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
percentage of participants | 22 | 32
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.308, Cochran-Mantel-Haenszel

4. Secondary Outcome: Annualized Flare Rate by British Isles Lupus Assessment Group (BILAG)-2004 Flare Index
Description: The BILAG-2004 index covers 86 questions item assessed across 9 organ systems. Each question is answered as 0-not present, 1-improving, 2- same, 3-worse, to 4-new.
  The BILAG-2004 index categorizes disease activity in each organ system into five different levels from A to E. Grade A represents requires disease-modifying treatment, Grade B represents mild, reversible problems requiring symptomatic therapy, Grade C indicates mild stable disease, and grade D implies no disease activity, but suggests the organ system had previously been affected. Grade E indicates no current or previous disease activity. Higher scores indicate more severe disease activity. Annualized flare rate is defined as the number of flares observed during the treatment period divided by the flare exposure time in days multiplied by 365.25.
Time Frame: From Baseline to Day 169
Population: mITT includes all randomized participants who received any amount of study drug and have completed at least one post-baseline disease assessment. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. Data was planned to be reported as LS Mean and Standard Error.
Measure: Least Squares Mean (Standard Error); unit: Flares per person-years
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
Flares per person-years | 3.27 (0.426) | 2.80 (0.426)
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.442, ANOVA

5. Secondary Outcome: Time-to-first Flare by BILAG-2004 Flare Index
Description: Time-to-first SLE flare is defined as the number of days from the administration of first dose to the first occurrence of flare. A flare was defined as having an adjudicated BILAG A or B score in any of the 8 organ systems during treatment. The BILAG disease activity index evaluates SLE activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease modifying treatment (prednisone greater than 20 mg daily or immunosuppressants); BILAG B: Disease less active than in "A", mild reversible problems requiring only symptomatic therapy such as antimalarials, NSAIDs, or prednisone less than 20 mg day; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved.
Time Frame: From Baseline to Day 169
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
days | 85.0 [57.0 to 112.0] | 113.0 [85.0 to 115.0]
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.788, Kaplan-Meier methods

6. Secondary Outcome: Percentage of Participants Achieving a Lupus Low Disease Activity State (LLDAS)
Description: The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. LLDAS was defined as SLE disease activity index (SLEDAI-2k <=4, with no activity in major organ systems (CNS, vascular, renal, cardiorespiratory and constitutional); where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0; No new features of lupus disease activity compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0; PGA (scale 0-3 higher scores = higher severity), <=1; current prednisolone (or equivalent) dose <=7.5 mg daily; and allowance for maintenance doses of immunosuppressive drugs and approved biological agents.
Time Frame: At Day 169
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
percentage of participants | 14 | 16
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.792, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Total Score
Description: SLEDAI-2K score is a disease activity score used to identify patients with more active disease at enrolment in study. Total score is defined as the sum of the weighted scores of each individual item within each organ system class. For each system organ with baseline score >0, improvement in SLEDAI-2K improvement is achieved by meeting all the following criteria:
  * Reduction in system organ scores among participants with baseline SLEDAI-2K scores greater than 0
  * No early discontinuation of study drug
  * No use of restricted medications beyond the protocol-allowed threshold before assessment
  SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: From Baseline to Day 169
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
score on a scale | -2.4 [-3.3 to -1.6] | -3.0 [-3.8 to -2.2]
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.302, Mixed models for repeated measures

8. Secondary Outcome: Cumulative Prednisone-equivalent Dose Use Through Day 169
Time Frame: From Baseline through Day 169
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligram (mg)
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 37 | 37
milligram (mg) | 1028.28 (183.729) | 854.59 (183.729)
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.506, ANOVA

9. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction In CLASI Activity Score In Participants With Baseline CLASI Activity Score ≥ 8
Description: CLASI is an validated measurement instrument for lupus erythematosus developed for use in clinical studies that consists of separate scores for the activity of the disease. CLASI Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and nonscarring alopecia. The total CLASI activity score ranges from 0-70, with higher scores indicating more severe skin disease.
Time Frame: From Baseline to Day 169
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
Number analyzed (Participants) | 10 | 11
percentage of participants | 30 | 45
Statistical Analysis 1: Comparison: ALPN-101 (Acazicolcept) vs Placebo; Test type: Superiority; p = 0.659, Fisher Exact

ADVERSE EVENTS:
Time Frame: Day 1 up to Safety follow-up (up to 28 weeks)
Description: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Arm/Group | ALPN-101 (Acazicolcept) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/38 | 2/38
Other Adverse Events (participants affected / at risk) | 18/38 | 16/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALPN-101 (Acazicolcept) (N=38) | Placebo (N=38)
Haemoglobin Decreased (Investigations) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALPN-101 (Acazicolcept) (N=38) | Placebo (N=38)
Aphthous Ulcer (Gastrointestinal disorders) | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
COVID-19 (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 0 | 2
Asthenia (General disorders) | 2 | 0
Influenza Like Illness (General disorders) | 0 | 2
Infusion Related Reaction (Immune system disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT04835441/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT04835441/SAP_001.pdf